CLINICAL TRIAL: NCT06203795
Title: Performance of Toxin Removal and Clotting Kinetics in Dialyzers
Brief Title: Dialysis Performance of the FX CorAL Membrane
Acronym: PATENCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0017 PATENCY
Record Dates: First submitted 2023-12-07; First posted 2024-01-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis Complication; Anticoagulants
Keywords: dialyzer fiber clotting
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hemodiafiltration with FX CorAL 800 dialyzer (Experimental): * Patients are dialyzed three consecutive dialysis sessions with an FX CorAL 800 dialyzer, starting on Saturday.
  * On Tuesday and Thursday, patients are dialyzed with only a quarter of their regular anticoagulation dose during 4 hours on Tuesday, and 3 hours on Thursday.
  * Blood is sampled from the arterial and venous blood line at different time points to determine concentrations of different uremic toxins and albumin
  Interventions: Other: Anticoagulation dosing; Other: Blood sampling; Other: Duration of the dialysis session; Device: Choice of the hemodialyzer
- Hemodiafiltration with FX 800 Cordiax dialyzer (Experimental): * Patients are dialyzed three consecutive dialysis sessions with an FX 800 Cordiax dialyzer, starting on Saturday.
  * On Tuesday and Thursday, patients are dialyzed with only a quarter of their regular anticoagulation dose during 4 hours on Tuesday, and 3 hours on Thursday.
  * Blood is sampled from the arterial and venous blood line at different time points to determine concentrations of different uremic toxins and albumin
  Interventions: Other: Anticoagulation dosing; Other: Blood sampling; Other: Duration of the dialysis session; Device: Choice of the hemodialyzer
- Hemodiafiltration with Solacea 19H dialyzer (Experimental): * Patients are dialyzed three consecutive dialysis sessions with a Solacea 19H dialyzer, starting on Saturday.
  * On Tuesday and Thursday, patients are dialyzed with only a quarter of their regular anticoagulation dose during 4 hours on Tuesday, and 3 hours on Thursday.
  * Blood is sampled from the arterial and venous blood line at different time points to determine concentrations of different uremic toxins and albumin
  Interventions: Other: Anticoagulation dosing; Other: Blood sampling; Other: Duration of the dialysis session; Device: Choice of the hemodialyzer
- Hemodiafiltration with Xevonta Hi-20 (Experimental): * Patients are dialyzed three consecutive dialysis sessions with a Xevonta Hi-20 dialyzer, starting on Saturday.
  * On Tuesday and Thursday, patients are dialyzed with only a quarter of their regular anticoagulation dose during 4 hours on Tuesday, and 3 hours on Thursday.
  * Blood is sampled from the arterial and venous blood line at different time points to determine concentrations of different uremic toxins and albumin
  Interventions: Other: Anticoagulation dosing; Other: Blood sampling; Other: Duration of the dialysis session; Device: Choice of the hemodialyzer

INTERVENTIONS:
Other: Anticoagulation dosing — Patients are dialyzed with only one quarter of their regular anticoagulation dose during the sessions on Tuesday and Thursday
Other: Blood sampling — Blood is sampled at start and at 10, 30, 60, 180, and 240 min after dialysis start for the 4 hours dialysis session, and at start and 10 and 180 min after dialysis start for the 3 hours dialysis session.
Other: Duration of the dialysis session — Patients have a washout with their regular dialysis duration on Saturday, a study session of 4 hours dialysis on Tuesday, and a study session of 3 hours dialysis on Thursday
Device: Choice of the hemodialyzer — Patients are dialyzed with one of the four dialyzers during the entire week, starting at Saturday (i.a. Saturday, Tuesday and Thursday). Block randomization is performed per two weeks. In week 1 and 2, patients are dialyzed with the FX CorAL 800 and the FX 800 Cordiax. In week 3 and 4 of the study, patients are dialyzed with the Solacea 19H and the Xevonta Hi20.

SUMMARY:
Anticoagulation remains an important issue in the setting of hemodialysis, and up till now there are some major points on which further research is needed. First, it is important to have a portfolio of the performance of different commercially available dialyzers with respect to fiber clotting. Second, to better estimate the impact of clotting on the overall dialysis performance, clotting kinetics during dialysis should be understood.

The aim of the present project is therefore to quantify the performance of the FX CorAL dialyzer (Fresenius Medical Care, Germany) in settings with reduced anticoagulation, and compare different performance outcomes (percent open fibers, solute removal rates) to those of other commercially available dialyzers. The different outcomes are related to the dialyzer extraction ratio and reduction ratio of small and middle molecules and albumin, the visual scoring of the dialyzer post dialysis, and the anticoagulation properties as assessed by fiber blocking in the dialyzer. Performance parameters at different time steps will allow to better understand clotting kinetics during dialysis.

DETAILED DESCRIPTION:
The FX CorAL is a polysulfone dialyzer with improved biocompatibility due to the increased polyvinylpyrrolidone (PVP) content on its blood side surface. Herewith, protein adsorption onto the membrane is lower, decreasing initiation of inflammation and suggesting less clotting problems.

The comPERFORM study already revealed the superiority of the FX CorAL 600 dialyzer versus the polysulfone-based Xevonta Hi15 (B. Braun, Germany) and the polyethersulfone-based Elisio 150H (Nipro, Japan) with respect to the clearance of Beta-2-Microglobulin at 60 min after dialysis start. Also the clearance of the larger toxin myoglobin was found superior in the FX CorAL, and removal rates, as calculated over the 240 min post dilution hemodiafiltration sessions, were superior in the FX CorAL for both middle molecules. Furthermore, albumin sieving properties of FX CorAL changed less over time than with the competitors.

Our group previously showed that here is a correlation between myoglobin dialyzer extraction and the percentage of open dialyzer fibers as quantified using the gold standard micro Computed Tomography (CT) scanning technique. However, previous data also suggested that fiber blocking during dialysis is not a linear process, but is rather accelerated during the second half of dialysis. Nevertheless, details about the kinetics of membrane and fiber clotting are still lacking. It can be hypothesized that the membrane pores and fibers in the FX CorAL have an improved tendency to remain open during the entire dialysis session, and that this will result in improved total solute removal, especially for middle molecules. Quantification of dialyzer fiber blocking using micro-CT scanning of dialyzer cross-sections, and this preferably after different durations of dialysis sessions, should be used to test this hypothesis. By including time points for performance measurements, like Extraction Ratio, with blood sampling e.g. at 10, 30, 60 min after dialysis start on the one hand, and at 180 and 240min, it might be possible to better understand clotting kinetics.

Polysulfone and polyethersulfone membranes have previously been associated with hypersensitivity reactions attributed to the use of additives such as PVP to enhance hydrophilic properties. In the FX CorAL however, the PVP is surface-stabilized and does not elute from the inner membrane surface. The Solacea dialyzer (Nipro, Japan), manufactured with an asymmetric triacetate (ATATM) membrane without hydrophilization agents, is also showing a lower risk of hypersensitivity, less decrease in platelets, and high permeability and filtration performance, and might be seen as a competitor for the FX CorAL.

Anticoagulation needs to be well-balanced to avoid an increased risk for bleeding complications on the one hand, and clotting of the extracorporeal circuit resulting in blood loss for the patient on the other hand. A high degree of fiber clotting in the early stage of the dialysis session might also result in decreased solute removal. More biocompatible membranes, such as FX CorAL and Solacea are theoretically less prone to coagulation problems during dialysis and could be used with decreased anticoagulation dose, reducing bleeding problems whilst still maintaining patency. The Solacea dialyzer showed maintained adequacy in conditions where systemic anticoagulation is contraindicated. Up till now, no studies to explore this in the FX CorAL have been performed.

The main questions the investigators want to answer with this study are:

1. How is fiber patency post dialysis in the FX CorAL versus competitors?
2. Can the FX CorAL be safely and adequately used in settings with reduced anticoagulation?
3. How is the time-dependent evolution of dialyzer extraction and clearance of small and middle molecules changing during the course of dialysis?
4. How is the time-dependent evolution of albumin loss?
5. How is the progression of membrane blockage and fiber blockage during the course of dialysis, i.e. during the last hour of a 4 hours dialysis session?

ELIGIBILITY:
Inclusion Criteria:

* stable chronic hemodialysis patient
* well functioning vascular access

Exclusion Criteria:

* known coagulation disorder
* active inflammation
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Fiber patency (i.e. number of open dialyzer fibers) in FX CorAL versus the competing dialyzers | 4 months
  Patients are dialyzed with four different dialyzers: FX CorAL 800, FX 800 Cordiax, Solacea 19H and Xevonta 20Hi
Calculation of dialyzer extraction in FX CorAL dialyzer in the setting of reduced anticoagulation | 4 months
  During the study dialysis sessions, patients only receive one quarter of their regular anticoagulation dose

SECONDARY OUTCOMES:
Time evolution of dialyzer extraction of uremic toxins and albumin | 4 months
  Blood is sampled at different time points to calculate extraction of different uremic toxins and albumin during dialysis
Time evolution of fiber patency during dialysis | 4 months
  Fiber patency is determined by micro Computed Tomography (CT) scanning after the dialysis session of 4 and 3 hours, respectively. By comparing the patency for those two sessions, we will learn about the progression of fiber clotting during 3 and 4 hours dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No